CLINICAL TRIAL: NCT06387043
Title: Comparison of the Effects of Balance Exercises Performed With Different Visual Stimuli in Individuals With Multiple Sclerosis
Brief Title: Effects of Balance Exercises Performed With Different Visual Stimuli
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Halic University (Other)
Collaborators: Fenerbahce University (Other); Biruni University (Other); Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gülsena Utku, Research Assistant, Halic University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MS and Balance
Record Dates: First submitted 2024-04-18; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; visual stimulus; balance; virtual reality; stroboscopic glasses; metaphoric imaginary
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Balance Games with Virtual Reality Glasses (Experimental): Individuals with MS in the first group will play balance games with virtual reality glasses for 15 minutes. Three different progressive games will be determined according to the functional level of the individual. Each game offers different gradually increasing difficulty levels and time options.
  Interventions: Other: Balance exercises with Virtual Reality Glasses
- Balance Exercises with Stroboscopic Glasses (Experimental): Individuals with MS in the second group will be given balance exercises with stroboscopic glasses for 15 minutes. Exercises will be selected in accordance with the functional level of the individual and will progress according to the individual's condition. In each session, 3-5 different exercises will be performed, taking into account the functional status of the individual.
  Interventions: Other: Balance Exercises with Stroboscopic Glasses
- Balance Exercises with Visual-Based Metaphor Training (Experimental): Individuals with MS in the third group will be given balance exercises simultaneously with metaphor training using various visuals for 15 minutes. The images will be projected on the screen in front of the individuals and the individuals will be given the command: "Imagine the movement you are doing as in the image." Meanwhile, reinforcers deemed necessary will be used by the researcher physiotherapist to increase the patient's participation and motivation. Static balance exercises in the program will be performed first on stable surfaces and then on unstable surfaces. In each session, 3-5 different exercises will be performed, taking into account the functional status of the individual. The difficulty levels of the exercises will progress by adjusting according to the functional status of the individual.
  Interventions: Other: Balance Exercises with Visual-Based Metaphor Training
- Traditional Balance Exercises (Active Comparator): Individuals with MS in the fourth group will be given balance exercises for 15 minutes under the supervision of a researcher physiotherapist. Exercises will be selected in accordance with the functional level of the individual and will progress according to the individual's condition. In each session, 3-5 different exercises will be performed, taking into account the functional status of the individual.
  Interventions: Other: Traditional Balance Exercises

INTERVENTIONS:
Other: Balance exercises with Virtual Reality Glasses — Balance exercises with Virtual Reality Glasses
  Arms: Balance Games with Virtual Reality Glasses
Other: Balance Exercises with Stroboscopic Glasses — Balance Exercises with Stroboscopic Glasses
  Arms: Balance Exercises with Stroboscopic Glasses
Other: Balance Exercises with Visual-Based Metaphor Training — Balance Exercises with Visual-Based Metaphor Training
  Arms: Balance Exercises with Visual-Based Metaphor Training
Other: Traditional Balance Exercises — Traditional Balance Exercises
  Arms: Traditional Balance Exercises

SUMMARY:
The study aims to examine the effects of balance exercises applied with different visual stimuli on individuals with MS.

DETAILED DESCRIPTION:
The study aims to examine the effects of balance exercises applied with virtual reality glasses, stroboscopic glasses, and visual-based metaphor imaginary on individuals with MS, on their balance functions, coordination skills, and quality of life, and to compare these exercises with both traditional balance exercises, and compare each of them on motor learning, based on their effects on representational areas in the brain, and balance.

ELIGIBILITY:
Inclusion Criteria:

* ages of 18-50
* diagnosis of MS by a neurologist according to McDonald 2017 criteria (Carroll, 2018)
* Being between 2.5 and 4.5 on the Expanded Disability Status Scale (EDSS)
* Not having had an attack in the last 3 months
* Absence of spasticity severe enough to affect treatment (spasticity in any joint of the upper extremity and lower extremity is <2 according to the Modified Ashworth Scale)
* Getting ≥ 24 points from the Standardized Mini Mental Test (SMMT)

Exclusion Criteria:

* hearing or vision problems
* pregnancy
* Having changed medication in the last 3 months and using medication containing the active ingredient Fampridine
* Participating or participating in a regular physiotherapy and rehabilitation program in the last 3 months
* other accompanying neurological, orthopedic or vestibular disorders
* an upper or lower extremity contracture that prevents exercises
* History of epileptic seizure, migraine or vertigo attack in the last 6 months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Functional Near Infrared Ray Spectroscopy (fNIRS) | Baseline and end of the 8th week
  Functional near-infrared spectroscopy is a device used to evaluate brain functions in the cerebral cortex. This device is an optical brain imaging method that measures the blood oxygenation level-dependent (BOLD) response of brain tissues. With this method, relative changes in regional brain oxygenation in the part thought to be associated with brain activation can be determined. In our study, Artinis Brite Lite® fNIRS systems will be used. The system consists of a wearable soft head and has 10 channels. In the evaluation procedure, a trial session will be conducted before the actual measurement, during which the subjects will be fitted with an fNIRS headset. The balance tasks to be evaluated will consist of right and left weight transfer, standing with two feet together, standing on one leg, tandem walking, turning from right to left/left to right, jumping in place and jumping over obstacles (Sathe et al., 2023).
Timed Up and Go Test | Baseline and end of the 8th week
  It is an assessment tool with strong evidence for its validity as a measure of functional mobility in individuals with MS ( Sebastiao et al., 2016 ).
Functional Reach Test | Baseline and end of the 8th week
  It is an easily applicable dynamic balance measurement technique that has features similar to functional movements. Distances below 15 cm have been found to be associated with an increased risk of falling (Weiner et al., 1992).
Berg Balance Scale | Baseline and end of the 8th week
  Berg Balance Scale is a scale that is widely used to evaluate balance disorders in multiple sclerosis patients (Berg et al., 1989), provides information about the patient's balance function, and is used to evaluate post-rehabilitation improvements (Gervasoni et al., 2016). The scale consists of 14 items for monitoring performance. Each item is scored between 0 and 4; A high score indicates good balance.
Timed 25 Step Walking Test | Baseline and end of the 8th week
  It will be used to evaluate the walking speed of individuals. In Z25YT, which evaluates lower extremity function, patients are asked to walk a distance of 7.62 m as quickly as possible, but without running and safely, and the completion time is recorded in seconds.

SECONDARY OUTCOMES:
Lower Extremity Motor Coordination Test | Baseline and end of the 8th week
  This test was developed by Desrosiers et al. to evaluate the lower extremity motor coordination skills of patients with a history of stroke, low back pain and surgery. Developed by. The test begins with the individual sitting on a chair with the knees and ankles at a 90-degree angle. Two red targets with a diameter of 6 cm are placed in front of it, distally and proximally, on a 55x50x0.4 cm mat, with 19 specific localization dimensions. The individual is asked to touch the target closest to the big toe as quickly and smoothly as possible. The number of movements made repetitively, smoothly and as fast as possible within 20 seconds is recorded (Desrosiers et al., 2005).
Fatigue Severity Scale | Baseline and end of the 8th week
  It is a scale consisting of 9 questions that evaluates fatigue. Each item is scored between 0 and 7. The total score is calculated by taking the arithmetic average of the scores. A score <4 is interpreted as no fatigue, and a score ≥4 as fatigue (Whitehead, 2009). The Turkish validity and reliability study of the scale was conducted by Armutlu et al., (Armutlu et al., 2007).
Quality of Life in Multiple Sclerosis Patients | Baseline and end of the 8th week
  Multiple Sclerosis Quality of Life Scale-54 was developed in 1995 by Vickrey et al. It was developed by (Vickrey et al., 1995); Turkish validity and reliability study by İdiman et al. Made by. The scale examines individuals' health-related quality of life levels with Likert-type scoring in a total of 54 questions prepared specifically for MS disease. Scoring varies between 0-100, with a higher score indicating a better quality of life (İdiman et al., 2006).

CONTACTS AND LOCATIONS:
Overall Officials: GÜLSENA UTKU UMUT, Principal Investigator — HALİÇ UNİVERSİTY
Locations (1):
- Haliç University, Istanbul, Eyüpsultan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided